CLINICAL TRIAL: NCT05726357
Title: Pulpotomy vs Root Canal Treatment for Teeth With Symptomatic Irreversible Pulpitis: A Randomised Control Trial
Brief Title: Pulpotomy vs Root Canal Treatment for Teeth With Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, shehabeldin saber, Professor, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FD BUE REC 22-034
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Pulpitis - Irreversible
Keywords: vital pulp therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard root canal treatment (Active Comparator): standard root canal treatment
  Interventions: Procedure: vital pulp therapy
- Pulpotomy (Active Comparator): vital pulp therapy
  Interventions: Procedure: vital pulp therapy

INTERVENTIONS:
Procedure: vital pulp therapy — removal of the coronal pulp followed by placing a biocompatible material to preserve the vitality of the radicular pulp

SUMMARY:
high-quality evidence is needed to add to current knowledge and also assess the long-term outcomes for full/complete pulpotomy after carious pulpal exposure in patients with signs and symptoms indicative of irreversible pulpitis

ELIGIBILITY:
Inclusion Criteria:

* a mature permanent tooth
* symptoms indicative of IRP
* responsive to cold and EPT sensibility testing
* restorable and can be adequately isolated during treatment
* One tooth (molar or premolar) per patient.

Exclusion Criteria:

* active periodontal disease
* complex medical histories
* unable to consent
* pregnant or breast-feeding
* excessive bleeding that cannot be controlled

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
pain score | day 3 post treatment
  score by a numeric rating scale from 1(minimum pain) to 100 (maximum pain)

SECONDARY OUTCOMES:
pain score | 6 months post treatment
  score by a numeric rating scale from 1(minimum pain) to 100 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: shehabeldin Saber, Principal Investigator — Professor of Endodontics
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not to be shared